CLINICAL TRIAL: NCT01391780
Title: Pelvic Floor Muscle Evaluation in Women With Stress Urinary and Urgency Urinary Incontinence. A Prospective Trial
Brief Title: Pelvic Floor Muscle Evaluation in Women With Stress Urinary and Urgency Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Prof. Trajano Sardenberg, Ethical Research Committee
Other Study IDs: 2011
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2011-03

CONDITIONS: Urinary Incontinence, Stress; Urge Incontinence
Keywords: pelvic floor evaluation,; women,; stress urinary incontinence;; urgency urinary incontinence.
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients with stress urinary incontinence
- Group 2: Patients with urgency urinary incontinence.

SUMMARY:
Aims: To assess pelvic floor muscle (PFM) strength in women with stress urinary incontinence (SUI) and urgency urinary incontinence (UUI).

Methods: 51 women were prospectively divided into two groups, according to the symptoms as SUI (G1 = 22) or UUI (G2 = 29). Demographic data, such as number of Pads/ 24 hours, number of micturitions/ 24 hours and nocturia, delay time of urgent void (i.e., the time period for which an urgent void could be voluntarily postponed), number of parity and vaginal deliveries were obtained using a clinical questionnaire. Objective urine loss was evaluated by 60-min Pad Test. Subjective [urine stream interruption test (UST), visual survey of perineal contraction and transvaginal digital palpation] and objective (vaginal manometry) evaluations of PFM were performed in all patients.

ELIGIBILITY:
Inclusion Criteria:

* presence of stress urinary or urgency incontinence

Exclusion Criteria:

* neurological diseases
* previous pelvic surgeries
* diabetes
* cognitive difficulties
* vaginal and urinary infection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was established considering a significance level of 5%, the test power of 80%, and the estimated error of 10%. According to these results and considering the range between percentages of answers as the casual error, each group was established with approximately 20 participants.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 1997-03; Study Completion 1998-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: João L. Amaro, PhD, MD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- São Paulo State University - Medical School of Botucatu, Botucatu, São Paulo, Brazil